CLINICAL TRIAL: NCT01165593
Title: Measurement of Left and Right Atria From CT Scans of Cardiac Rhythm Disorder Cases
Status: Completed | Type: Observational
Sponsor: Kardium Inc. (Industry)
Collaborators: St. Paul's Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: H10-01337
Record Dates: First submitted 2010-07-16; First posted 2010-07-20 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with atrial fibrillation: Patients with atrial fibrillation who have received a cardiac CT scan as part of normal care prior to catheter-based treatment of atrial fibrillation.
  Interventions: Other: There is no intervention that is a part of this study.

INTERVENTIONS:
Other: There is no intervention that is a part of this study. — There is no intervention that is a part of this study. Imaging data is gathered as part of normal care.

SUMMARY:
The purpose of this study is to gather information about the size and shape of patients' hearts in order to design a device.

DETAILED DESCRIPTION:
Correct device design depends on getting good information about the shape and size of the different parts of the heart. Measurements from computed tomography images of hearts will be studied. By looking at measurements from a wide range of patients, an understanding of the differences in the size and shape of the heart chambers will be gained.

ELIGIBILITY:
Inclusion Criteria:

* Patients deemed suitable for treatment of atrial fibrillation by catheter-based ablation who have received cardiac CT imaging as part of normal care.

Exclusion Criteria:

* Patients who have not received cardiac CT imaging as part or normal care.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with atrial fibrillation who are deemed suitable for treatment of atrial fibrillation by catheter-based ablation.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2010-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
LA size measurements | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: John A. Yeung-Lai-Wah, MD, Principal Investigator — St' Paul's Hospital Electrophysiology (Providence Health Care)
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada